CLINICAL TRIAL: NCT02799108
Title: Analysis of Lateralization of Language in Epileptic Children by Near-infrared Spectroscopy (NIRS)
Acronym: LANGLAT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: inclusion difficulty
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AOL11-DR-WALLOIS
Record Dates: First submitted 2016-06-09; First posted 2016-06-14 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Epilepsy
Keywords: children; language; NIRS
MeSH Terms: conditions — Epilepsy; Language | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- patients (Experimental): children with drug-resistant partial epilepsy, in whom preoperative assessment is indicated
  Interventions: Device: NIRS; Device: fMRI

INTERVENTIONS:
Device: NIRS — High-resolution EEG-fNIRS recording lasting a maximum of 30 minutes by using expressive and receptive language paradigms
Device: fMRI — fMRI acquisition under the same stimulation conditions

SUMMARY:
Recent data published by various laboratories as well as our preliminary data tend to prove that near-infrared spectroscopy can be used to determine the lateralization of language as part of the preoperative assessment for drug-resistant epilepsy. The reference test used up until very recently was the Wada test, which consisted of injecting an anaesthetic (generally amobarbital sodium) into one of the internal carotid arteries (right or left) in order to determine the predominant cerebral hemisphere for language. This invasive test has been progressively replaced by fMRI, which is nevertheless difficult to perform in children under the age of 7 years. NIRS therefore appears to be a useful alternative, which, in contrast with fMRI, can be easily repeated and allows simple investigation of the various facets of language (e.g. expressive, receptive). In the GRAMFC unit, the investigators have acquired a unique know-how in the field of high-resolution NIRS, both in epilepsy and in the development of language structures.

ELIGIBILITY:
Inclusion Criteria:

* children with drug-resistant partial epilepsy, in whom preoperative assessment is indicated.

Exclusion Criteria:

* All children with severe congenital malformation
* Any refusal of a parent or child
* Any child with generalized epilepsy or diffuse interictal spikes
* Any child with a serious deterioration in the general condition and vital functions
* Any child with dermatitis of the face or scalp
* Children under 6 years

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2012-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
lateralization index | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Fabrince WALLOIS, MD,PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France